CLINICAL TRIAL: NCT04040231
Title: Combining a WT1 Cancer Vaccine (Galinpepimut-S) With Checkpoint Inhibition (Nivolumab) in Patients With WT1-Expressing Malignant Pleural Mesothelioma: A Phase I Study
Brief Title: Using a Targeted Cancer Vaccine (Galinpepimut-S) With Immunotherapy (Nivolumab) in Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-654
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Mesothelioma; Pleural Mesothelioma; Wilms Tumor
Keywords: Mesothelioma; Pleural Mesothelioma; Wilms Tumor Protein 1; WT1; galinpepimut-S; Montanide; Nivolumab; Phase I; 17-654; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant; Wilms Tumor | interventions — Nivolumab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Malignant Pleural Mesothelioma (MPM) (Experimental): Participants with previously treated Malignant Pleural Mesothelioma/MPM
  Interventions: Biological: Galinpepimut-S; Drug: Nivolumab; Biological: Sargramostim

INTERVENTIONS:
Biological: Galinpepimut-S — Galinpepimut-S will be administered alone on weeks 0 and 2. Participants will receive the galinpepimut-S vaccine and nivolumab over 16 weeks in the initial treatment phase.
Drug: Nivolumab — Participants will receive nivolumab and the galinpepimut-S vaccine over 16 weeks in the initial treatment phase.
Biological: Sargramostim — All participants will receive Sargramostim (GM-CSF) 70 mcg injected subcutaneously on days 0 and -2 of each cycle
  Other Names: GM-CSF

SUMMARY:
The purpose of this study is to test whether it is safe to give Galinpepimut-S and Nivolumab together in patients with mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Karnofsky performance status >/= 70%
* Pathologic diagnosis of malignant pleural mesothelioma at MSK
* Positive immunohistochemical staining for WT-1 within 60 days of treatment start
* Patients must have received at least one prior course of pemetrexed-based chemotherapy
* Patients of childbearing potential must have a negative serum pregnancy test within 24 hours of receiving the first treatment on the study (if female) and must be practicing an effective form of birth control for the entire duration of treatment (both females and males)
* Has received and progressed or are refractory to pemetrexed based chemotherapy
* Measurable or evaluable disease
* Biochemical parameters: Total bilirubin < 1.5 mg/dl, AST and ALT < 3.0 x upper limits of normal, Creatinine < 1.5 x upper limits of normal

Exclusion Criteria:

* Pregnant or lactating women
* Prior receipt of checkpoint inhibition
* Patients with known active hepatitis B or known active hepatitis C virus
* Patients with a serious unstable medical illness or another active cancer
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Autoimmune disease requiring treatment with systemic steroids in the past 2 years
* Current use of systemic corticosteroids at doses greater than prednisone 10 mg daily or the equivalent
* Patients with active pneumonitis
* Hematologic parameters: Absolute neutrophil count >/= 1000/mcL
* Platelet count <100,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | up to 24 months
  A dose will be considered tolerable if there are no more than 2 out of 10 participants with dose limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Offin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org